CLINICAL TRIAL: NCT04717479
Title: A Scalable Model for Promoting Functioning and Well-Being Among Older Adults With Mild Cognitive Impairment Via Meaningful Social Interactions: Project SPEAK!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John Piette, Professor of Health Behavior and Health Education, and of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R21AG066644 (NIH); 5R21AG066644-02 (NIH)
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Participants will be paired with an English language learner and engage in 8 weeks, 1 hour videoconferencing sessions.
  Interventions: Other: Intervention (videoconferencing)
- Wait-list Control (Other): Participants will wait 8 weeks and then they will be paired with an English language learner and engage in 8 weeks, 1 hour videoconferencing sessions.
  Interventions: Other: Intervention (videoconferencing)

INTERVENTIONS:
Other: Intervention (videoconferencing) — 1 hour videoconferencing sessions over 8 weeks with an English language learner partner.

SUMMARY:
The goal of this study is to refine and test a strategy for engaging older adults with symptoms of SCD/MCI (subjective cognitive decline/mild cognitive impairment) as volunteers to help English language learners (ELLs) who live in the US improve their speaking skills via structured conversations using videoconferencing.

DETAILED DESCRIPTION:
Aim 1: Conduct a user-centered design process to refine the SPEAK! training protocols for older adults with symptoms of SCD/MCI and ELLs, and the materials that will support productive engaging English conversation practice.

Aim 2: Conduct a randomized, wait-list controlled trial of 8 weeks of SPEAK! participation, using a variety of recruitment sources, in order to evaluate our capacity to recruit, implement the intervention, and retain older adults with symptoms of SCD/MCI in sufficient numbers for a subsequent randomized-controlled trial evaluating the intervention's impact on participants' psychological well-being, mood, and cognitive functioning.

Aim 3: Using mixed methods, evaluate the communication process between older adults with symptoms of SCD/MCI and ELLs including factors that contribute to satisfaction of both parties, engagement in planned contacts, possible contributors to stress or dissatisfaction, and perceptions among older adults of being appreciated and effective. The investigators will also estimate variances for key outcome variables and conduct exploratory analyses of intervention-control differences in participants' perceptions of their wellbeing, mood, and cognitive functioning.

ELIGIBILITY:
Mild Cognitive Impairment participant --

Inclusion Criteria:

* 55+ years of age, fluent speakers of English of any race/ethnicity, and be able to participate in a videoconference via a smartphone, tablet laptop, or desktop computer in their home or referring organization using a widely accessible, no cost videoconferencing platform.

Exclusion Criteria:

* Participants will be ineligible if they have a history of stroke or traumatic brain injury, bipolar disorder, schizophrenia, or current alcohol or drug abuse/dependence, that would affect their ability to participate in the study; MoCA score <12.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Piette, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, North Campus Research Complex, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Goal of recruiting 44 pairs into the waitlist trial for AIMS 2-3.
Period: Overall Study
Arm/Group | Intervention | Wait-list Control
Started | 41 (41 individuals -- 22 MCIs and 19 ELLs) | 39 (39 individuals -- 22 MCIs and 17 ELLs)
Completed | 34 (34 individuals -- 17 MCIs and 17 ELLs) | 35 (35 individuals -- 21 MCIs and 14 ELLs)
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Wait-list Control | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Information was not obtained for one ELL participant
  years
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): number analyzed (Participants) | 22 | 22 | 44
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline) | 70 (9.49) | 71 (8.06) | 71 (8.82)
    ELL (English Language Learner): number analyzed (Participants) | 19 | 17 | 36
    ELL (English Language Learner) | 41 (9.73) | 43 (9.07) | 42 (9.32)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Overall population described in two groups: MCI/SCD participants and ELL participants
  Participants
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): number analyzed (Participants) | 22 | 22 | 44
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Female | 12 | 16 | 28
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Male | 10 | 6 | 16
    ELL (English Language Learner): number analyzed (Participants) | 19 | 17 | 36
    ELL (English Language Learner): Female | 15 | 13 | 28
    ELL (English Language Learner): Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall population described in two groups: MCI/SCD participants and ELL participants
  Participants
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): number analyzed (Participants) | 22 | 22 | 44
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Hispanic or Latino | 0 | 0 | 0
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Not Hispanic or Latino | 22 | 22 | 44
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Unknown or Not Reported | 0 | 0 | 0
    ELL (English Language Learner): number analyzed (Participants) | 19 | 17 | 36
    ELL (English Language Learner): Hispanic or Latino | 11 | 12 | 23
    ELL (English Language Learner): Not Hispanic or Latino | 8 | 5 | 13
    ELL (English Language Learner): Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall population analyzed in 2 groups: MCI/SCD participants and ELL participants
  Participants
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): number analyzed (Participants) | 22 | 22 | 44
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): American Indian or Alaska Native | 0 | 0 | 0
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Asian | 2 | 0 | 2
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Black or African American | 4 | 7 | 11
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): White | 16 | 15 | 31
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): More than one race | 0 | 0 | 0
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Unknown or Not Reported | 0 | 0 | 0
    ELL (English Language Learner): number analyzed (Participants) | 19 | 17 | 36
    ELL (English Language Learner): American Indian or Alaska Native | 0 | 0 | 0
    ELL (English Language Learner): Asian | 4 | 4 | 8
    ELL (English Language Learner): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    ELL (English Language Learner): Black or African American | 1 | 1 | 2
    ELL (English Language Learner): White | 9 | 10 | 19
    ELL (English Language Learner): More than one race | 3 | 0 | 3
    ELL (English Language Learner): Unknown or Not Reported | 2 | 2 | 4
Highest Degree of Completed Education [Count of Participants; unit: Participants] — Population: Overall population analyzed in 2 groups: MCI/SCD participants and ELL participants
  Participants
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): number analyzed (Participants) | 22 | 22 | 44
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): 8th grade or less | 0 | 0 | 0
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Some high school,but did not graduate | 0 | 0 | 0
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): High school graduate or GED | 1 | 2 | 3
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Some college or two-year college degree | 5 | 3 | 8
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): Four-year college graduate | 6 | 9 | 15
    MCI/SCD (Older adults with mild cognitive impairment/subjective cognitive decline): More than four-year college degree | 10 | 8 | 18
    ELL (English Language Learner): number analyzed (Participants) | 19 | 17 | 36
    ELL (English Language Learner): 8th grade or less | 0 | 0 | 0
    ELL (English Language Learner): Some high school,but did not graduate | 0 | 0 | 0
    ELL (English Language Learner): High school graduate or GED | 0 | 0 | 0
    ELL (English Language Learner): Some college or two-year college degree | 2 | 1 | 3
    ELL (English Language Learner): Four-year college graduate | 7 | 4 | 11
    ELL (English Language Learner): More than four-year college degree | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of MCI/SCD (Mild Cognitive Impairment/Subjective Cognitive Decline) Participants Recruited Within the First Six Months
Description: The primary aim for Phase 2 of the study was to demonstrate the feasibility of recruiting and consenting a minimum of 35 older adults with MCI/SCD (mild cognitive impairment/subjective cognitive decline) within the first six months.
Time Frame: Baseline (Up to approximately 1 hour and 15 minutes over the course of two meetings).
Population: The overall number of participants analyzed refers to the 50 participants that were screened in the first 6 months, from which 35 participants were enrolled in the first 6 months.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Overall participant recruitment of MCI/SCD (older adults with mild cognitive impairment/subjective cognitive decline) arm of the study within the first six months.
Arm/Group | Overall
Number analyzed (Participants) | 50
Participants | 35

2. Other Pre Specified Outcome: Psychological Wellbeing Scale (PWB)
Description: The Psychological Wellbeing Scale (PWB) is a validated measure shown to be sensitive to intervention effects. This is a 6 point scale where the minimum is 1 (strongly disagree) and maximum is 6 (strongly agree). Higher scores reflect higher wellbeing.
Time Frame: Baseline and follow-up collected after the 8-week intervention time period.
Reporting Status: Not Posted

3. Other Pre Specified Outcome: UCLA Revised Loneliness Scale
Description: This is a validated measure of loneliness with an alpha reliability of .94. This is a 4 point scale from 1=never to 4=always (minimum is 1 maximum is 4). Positively worded questions will be reverse-coded so that higher scores mean more loneliness.
Time Frame: Baseline and follow-up collected after the 8-week intervention time period.
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Geriatric Depression Scale
Description: The Geriatric Depression Scale is a measure of depressive symptoms specifically designed for older adults. The 30 point scale has a minimum of 0 points to maximum 30 points. Higher scores reflect greater depression.
Time Frame: Baseline and follow-up collected after the 8-week intervention time period.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months during recruitment and delivery of the intervention.
Description: Reviewed by staff during our weekly meetings. Same definition as in clinicaltrials.gov.
  All serious events were unrelated to the study.
Arm/Group | Intervention | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 2/41 | 1/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=41) | Wait-list Control (N=39)
Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Car accident injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT04717479/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT04717479/ICF_000.pdf